CLINICAL TRIAL: NCT04878497
Title: Prospective Monitoring of Non-Vitamin K Oral Anticoagulants in Older Adults With Atrial Fibrillation and Frailty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Dae Hyun Kim, MD, MPH, ScD, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2019P000110-NOAC
Record Dates: First submitted 2021-04-22; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation; Frailty; Anticoagulant-induced Bleeding; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Frailty; Stroke | interventions — Warfarin; Dabigatran; Rivaroxaban; apixaban; edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Warfarin: New users of warfarin
  Interventions: Drug: Warfarin
- Dabigatran: New users of dabigatran
  Interventions: Drug: Dabigatran
- Rivaroxaban: New users of rivaroxaban
  Interventions: Drug: Rivaroxaban
- Apixaban: New users of apixaban
  Interventions: Drug: Apixaban
- Edoxaban: New users of edoxaban
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Warfarin — Initiation of warfarin, identified using prescription fill in pharmacy claims
  Groups: Warfarin
Drug: Dabigatran — Initiation of dabigatran, identified using prescription fill in pharmacy claims
  Groups: Dabigatran
Drug: Rivaroxaban — Initiation of rivaroxaban, identified using prescription fill in pharmacy claims
  Groups: Rivaroxaban
Drug: Apixaban — Initiation of apixaban, identified using prescription fill in pharmacy claims
  Groups: Apixaban
Drug: Edoxaban — Initiation of edoxaban, identified using prescription fill in pharmacy claims
  Groups: Edoxaban

SUMMARY:
The objective of this study is to establish a near-real-time prospective monitoring program in Medicare, Optum and MarketScan Research data to evaluate the benefit of new cardiovascular disease (CVD) drugs for older adults with frailty. Prospective monitoring program seeks to find early effectiveness and safety signals of new drugs by updating the analysis at regular intervals as new Medicare data become available. This study specifically aims to emulate a prospective surveillance of the effectiveness and safety of non-vitamin K oral anticoagulants (NOAC) vs. a comparator, warfarin, in older adults with atrial fibrillation and different frailty status. This program will be enhanced by incorporating a novel claims-based frailty index, which has been shown useful in assessing how the benefits and harms of drug therapy vary by frailty.

DETAILED DESCRIPTION:
Data sources of use for this study are: Medicare Database, Optum Database, and MarketScan Research Database. All data from years 2013-2020 (available data may vary depending on the database) will be analyzed in the study.

This study follows a sequential cohort monitoring design. The monitoring analysis will include 1) retrospective analysis of available data (2013-2018) at the time of first analysis (April 2021) and 2) prospective analysis of new data (2019-2020) as they become available to the researchers. Within each database and by frailty status (frail vs non-frail), the investigators will emulate annual updating of data by creating a propensity score (PS)-matched cohort of new users every 1-year interval. Each sequential cohort will be followed for development of the outcomes of interest. At the end of each interval, time-to-event data from all sequential cohorts will be pooled for outcome analysis. The surveillance will be performed by frailty status (frail vs non-frail) at the time of drug initiation.

ELIGIBILITY:
Inclusion Criteria:

* Initiation of a NOAC or warfarin (day 0 is the initiation day)
* Continuous enrollment in medical and drug insurance in [-183, 0] days
* Diagnosis of AF in [-183, 0] days
* CHA2DS2-VASc score ≥2 (moderate or high risk for stroke)
* No prior use of NOAC or warfarin in [-183, -1] days
* No recent hospitalization for stroke or major bleeding in [-60, 0] days
* No recent nursing facility stay in [-60, 0] days

Exclusion Criteria:

* Contraindication to either drug in [-183, 0] days
* Valvular heart disease or mechanical heart valve in [-183, 0] days
* Intracranial or retroperitoneal hemorrhage in [-183, 0] days
* Chronic kidney disease stage V, end-stage renal disease, or dialysis in [-183, 0] days
* Other indications for anticoagulation therapy in [-183, 0] days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Study population includes older patients with non-valvular AF who initiates warfarin or a NOAC.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with composite events of stroke or systemic embolism | January 2013 - December 2020 (after drug initiation)
  Stroke OR systemic embolism, identified by relevant diagnoses in the claims data
Number of patients with major bleeding | January 2013 - December 2020 (after drug initiation)
  Major bleeding, identified by relevant diagnoses in the claims data

SECONDARY OUTCOMES:
Number of patients with all-cause mortality | January 2013 - December 2020 (after drug initiation)
  All-cause mortality is defined by the National Death Index file or vital status information in the claims data.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Kim, MD, MPH, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT04878497/Prot_SAP_000.pdf